CLINICAL TRIAL: NCT01228604
Title: COST-EFFECTIVENESS STUDY OF THE TREATMENT OF ATTENTION DEFICIT/HYPERACTIVITY DISORDER IN BRAZIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100021
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: open label; Ritalin®; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

ARMS (1):
- Methylphenidate (Experimental)
  Interventions: Drug: methylphenidate (Ritalin®)

INTERVENTIONS:
Drug: methylphenidate (Ritalin®) — The scheme provides for initial dose of 0.3 mg / kg / day, with an average dose of 1mg/kg/day. The increases will be made considering the presentation of the drug (10mg), which allows increments of 5mg or 10mg, which will be made in clinical review, as the clinical symptoms, including increasing the dose until there is more room for improvement or there is presence of significant adverse effects, all the patients with indication of treatment will be assessed before the use of medication, 15 days, 30 days, 3 and 6 months after the start,

SUMMARY:
This study is an open-label, 6 month trial, of immediate release methylphenidate (MPH-IR) for children with ADHD aimed at assessing whether the observable behavioral changes seen during treatment are associated with potentially more stable underlying modifications in brain functioning (resting-state functional connectivity). Additionally, we will also be looking at treatment effects on neuropsychological processes and reading skills. This information will contribute to the first Brazilian study assessing the cost-effectiveness of the treatment of ADHD. Children with ADHD will be compared to a sample of sex and age-matched sample of typically developing children.

ELIGIBILITY:
Inclusion Criteria:

The study will include 20 boys aged 8 to 10 years old, regularly enrolled in local schools and directed to the research through advertisement in the media, contact with schools or directly referred to the Attention Deficit/Hyperactivity Program (ProDAH/HCPA) by primary care services for assessment and treatment. Only children with a primary diagnosis of ADHD or with the comorbidity ADHD + reading disorder or ADHD + ODD will be included. Only drug-naïve subjects will be apt to participate in the study.

Exclusion Criteria:

Children who fit into one or more of the following conditions will not be considered eligible to take part in the study: (1) they are outside the age range specified; (2) they are not regularly enrolled and attending school; (3) they have a history of prior or current treatment with psychoactive drugs or psychotherapy; (4) they are mentally retarded (Overall IQ<80); (5) they have a main diagnosis differing from ADHD, including children with other psychiatric or neurological diagnoses

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Resting-state functional connectivity | After 6 months
  After 6 months of treatment, participants will perform a second fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil